CLINICAL TRIAL: NCT01421381
Title: A Single Visit, Observational, Follow-up Study of Patients With Leber's Hereditary Optic Neuropathy Following Participation in SNT-II-003 Trial
Brief Title: RHODOS Follow-up Single-visit Study
Acronym: RHODOS-OFU
Status: Completed | Type: Observational
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNT-II-003-OFU
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Leber's Hereditary Optic Neuropathy
Keywords: leber's hereditary optic neuropathy; idebenone
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study aims to evaluate the current visual acuity of SNT-II-003 participants and compare this with the last visit from the SNT-II-003 study.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in study SNT-II-003

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who participated in study SNT-II-003
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
logMAR visual acuity | measure taken at the single study visit (Week 24)
  Change in best logMAR visual acuity (Best Acuity) compared to Visit 2/Baseline and Visit 5/Week 24 or last treatment visit of SNT-II-003

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chinnery, MD, Principal Investigator — Clinical Research Facility
Locations (3):
- Hôpital Notre-Dame (CHUM), Montreal, Quebec, Canada
- Friedrich Baur Institut Neurologische Klinik und Poliklinik, München, Germany
- Biomedical Research Centre, The Medical School, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Background] Klopstock T, Yu-Wai-Man P, Dimitriadis K, Rouleau J, Heck S, Bailie M, Atawan A, Chattopadhyay S, Schubert M, Garip A, Kernt M, Petraki D, Rummey C, Leinonen M, Metz G, Griffiths PG, Meier T, Chinnery PF. A randomized placebo-controlled trial of idebenone in Leber's hereditary optic neuropathy. Brain. 2011 Sep;134(Pt 9):2677-86. doi: 10.1093/brain/awr170. Epub 2011 Jul 25. PMID 21788663
- [Result] Klopstock T, Metz G, Yu-Wai-Man P, Buchner B, Gallenmuller C, Bailie M, Nwali N, Griffiths PG, von Livonius B, Reznicek L, Rouleau J, Coppard N, Meier T, Chinnery PF. Persistence of the treatment effect of idebenone in Leber's hereditary optic neuropathy. Brain. 2013 Feb;136(Pt 2):e230. doi: 10.1093/brain/aws279. Epub 2013 Feb 6. No abstract available. PMID 23388409